CLINICAL TRIAL: NCT03205592
Title: Ultrasound Assessment of Residual Gastric Content in Critically Ill Patients
Acronym: GastrICU
Status: Completed | Type: Observational
Sponsor: Hôpital Edouard Herriot (Other)
Responsible Party: Principal Investigator, Lionel Bouvet, Principal investigator, Hôpital Edouard Herriot
Other Study IDs: L16-174
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Critically Ill Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasound examination of the antrum — Ultrasound assessment of gastric content will be performed : prior to suction of gastric content through a gastric tube (method to assess the residual gastric content volume), after this suctioning of gastric content, then after reinjection of the content suctioned into the stomach (max 250 ml) and 1h30 later

SUMMARY:
This prospective observational study aims to assess whether ultrasound assessment of gastric content may be useful for the monitoring of the gastric residual content in critically ill patients

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients under mechanical ventilation and enteral feeding through a gastric tube since >48 h

Exclusion Criteria:

* Digestive hemorrhage Contra-indication to prokinetic drugs Enteral feeding through jejunostomy or gastrostomy Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients hospitalized in 3 critical care units (Groupement hospitalier Sud Lyon, Saint Etienne, Marseille)
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2018-05-04 (Actual); Study Completion 2018-05-04 (Actual)

PRIMARY OUTCOMES:
change in antral cross sectional area measured by ultrasonography after suctioning gastric volume | prior to and immediately after suctioning of gastric content volume through a gastric tube
  Ultrasound measurement of antral area and qualitative assessment
Change in antral area after administration of prokinetic drug | Ultrasound assessment of gastric content after reinjection of suctioned gastric content and 1h30 later (1 h after the end of the infusion of prokinetic drug)
  If aspirated gastric content volume was > 250 ml, only 250 ml will be reinjected into the stomach and a prokientic drug will be administered (current protocol in our units). Antral area will be measured prior to and 90 min after the start of the infusion

CONTACTS AND LOCATIONS:
Overall Officials: Lionel BOUVET, MD PhD, Principal Investigator — Hospices Civils de Lyon
Locations (3):
- France (3):
  - Hôpital Nord, Marseille
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Saint Etienne, Saint-Etienne

REFERENCES:
- [Derived] Bouvet L, Zieleskiewicz L, Loubradou E, Alain A, Morel J, Argaud L, Chassard D, Leone M, Allaouchiche B; AzuRea CAR'Echo collaborative networks. Reliability of gastric suctioning compared with ultrasound assessment of residual gastric volume: a prospective multicentre cohort study. Anaesthesia. 2020 Mar;75(3):323-330. doi: 10.1111/anae.14915. Epub 2019 Dec 4. PMID 31802485